CLINICAL TRIAL: NCT00170456
Title: A Double-Blind, Parallel-Group Study of the Safety, Tolerability and Immunogenicity of a Range of Doses and Dosing Schedules of Recombinant (rPA Based) Anthrax Vaccine in Healthy Subjects
Brief Title: Phase II Study of Range and Schedule of rPA Doses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmAthene UK Limited (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 05-0003; QGUY/2004/AV-rPA/-01
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2008-09-15 (Estimated); Status verified 2008-09

CONDITIONS: Prevention of Bacillus Anthracis (Anthrax) Infection
Keywords: Anthrax vaccine
MeSH Terms: conditions — Anthrax; Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Low dose rPA vaccine regime 1
  Interventions: Biological: rPA vaccine containing alhydrogel
- 2 (Active Comparator): Low dose rPA vaccine regime 2
  Interventions: Biological: rPA vaccine containing alhydrogel
- 3 (Active Comparator): High dose rPA vaccine regime 1
  Interventions: Biological: rPA vaccine containing alhydrogel
- 4 (Active Comparator): High dose rPA vaccine regime 2
  Interventions: Biological: rPA vaccine containing alhydrogel

INTERVENTIONS:
Biological: rPA vaccine containing alhydrogel

SUMMARY:
This is a dose ranging study comparing different vaccine schedules of rPA vaccine for anthrax. Safety and the capability to induce an immune response will be evaluated.

DETAILED DESCRIPTION:
Anthrax is a zoonotic disease, occurring in wild and domestic mammals, caused by the spore forming bacterium Bacillus anthracis. Anthrax occurs in humans when they are exposed to infected animals, tissue from infected animals or when they are directly exposed to B. anthracis or its spores. In the USA, the annual incidence of human anthrax has declined. However, in the USA, shortly after September 11th 2001, there were 22 cases (18 confirmed) of inhaled and cutaneous anthrax infections that were related to contaminated mail. This is a double blind, parallel-group, dose ranging study of rPA anthrax vaccine. The subjects will be blinded as to which dose of rPA vaccine is administered. The primary objectives of this clinical trial are 1.) To evaluate the safety and tolerability associated with different primary immunization doses and schedules of rPA vaccine to enable determination of the optimum dose for future clinical trials and 2.) To evaluate the immunogenicity of different primary immunization doses and schedules of rPA vaccine to enable determination of the optimum schedule for future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females.
2. Aged between 18-55 years (inclusive).
3. A body mass index (BMI) of 18-35.
4. Signed informed consent, which includes information about the potential risks and effects of rPA.
5. A medical history without major organ pathology (e.g. cardiac, immunological, psychiatric, endocrine or neurological disorders, cancer or other wasting diseases - (adequately treated actinic keratosis, or basal cell carcinoma [BCC], or carcinoma in situ [CIS] of the cervix are permitted).
6. A female may be enrolled if one of the following criteria applies:

   Either If of child-bearing capacity then: A female is not pregnant or breast feeding AND is routinely using adequate injectable or transdermal (administered at the recommended frequency) or oral contraception (at a stable dose for at least three months prior to the first dose of vaccine) and will continue to do so during the study, augmenting this contraceptive measure with a barrier method OR is sexually abstinent OR is monogamous and has a partner who has had a vasectomy (>1 month previously) OR is using a commonly recognised copper and hormone implanted intrauterine device (IUD) such as TCu-380A, TCu-220C, MLCu-375, Nova-T or LNG-20. In addition, the subject must have a negative blood pregnancy test prior to enrolment into the study and negative urine pregnancy test pre-dose.

   Or A female is post menopausal (defined as a female with no menstrual cycle for at least 24 months and of menopausal age (>45 years).

   Or A female with no menstrual cycle for between 12 and 24 months and of menopausal age (>45 years) who has a negative blood pregnancy test prior to enrolment into the study and a negative urine pregnancy test pre-dose.

   Or A female has been surgically sterilised (confirmed by review of medical record).

   Or A female has had a total hysterectomy at least 3 months prior to the start of the study (confirmed by review of medical record).
7. A male may be enrolled if willing to use barrier methods of contraception and whose partner is using an acceptable form of contraception for 3 months post each dose.
8. Able to understand the informed consent form and other documents required to be read by the subject.

Exclusion Criteria:

1. Presence of any clinically significant medical condition as determined by the Investigator.
2. Medically significant hypersensitivity or idiosyncratic reaction related to any medical product including vaccines.
3. History or evidence of drug abuse.
4. Participation in a clinical study of an investigational vaccine within 3 months prior to the start of the study or an investigational drug product within 30 days prior to the start of the study.
5. Use of any prescription or non-prescription medication within 7 days prior to the first dosing with the exception of over-the-counter (OTC) antihistamine, non-steroidal anti-inflammatory drugs (NSAID), acetaminophen, OTC decongestants or oral/injectable/transdermal contraceptives. Any medication taken within 7 days of the first dosing will be recorded.
6. History or suspicion of inability to co-operate adequately.
7. Donation of blood or blood products for a period of 4 weeks prior to participation in the study.
8. Immunodeficiency or clinically active autoimmune disease.
9. Positive urine alcohol and drug screen for drugs of abuse (opiates, methadone, cocaine, amphetamines, cannabinoids, and barbiturates).
10. Positive test for human immunodeficiency virus (HIV), and/or hepatitis B and/or hepatitis C.
11. Vaccination(s) with a live vaccine in the previous 4 weeks or killed / inactivated vaccines in the previous 3 weeks.
12. Blood or plasma transfusions, or pooled gamma-globulin in the previous 3 months and need for blood or plasma transfusions during this study.
13. Received anthrax vaccine or anthrax immune globulin or been otherwise exposed to B. anthracis.
14. Clinically relevant abnormal findings on routine physical examination.
15. Clinically significant out-of-range laboratory tests at screening including: urinalysis, serum creatinine, lactate dehydrogenase (LDH), potassium, glucose, liver function tests (LFT); absolute neutrophil count, platelet count, white blood cell count, electrolytes, clotting and blood haemoglobin.
16. Twelve-lead ECG recording with clinically relevant signs of pathology and conduction disturbances as judged by the investigator.
17. Presence of tattoos that cover or partially cover the upper arm.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 415 (Actual)
Dates: Start 2005-03; Primary Completion 2007-01 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Safety of rPA vaccine

SECONDARY OUTCOMES:
Immunogenicity of rPA vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Mant, MD, Principal Investigator — GDRU, London, UK
Locations (2):
- United Kingdom (2):
  - GDRU, Quintiles Ltd, London
  - Simbec Research Limited, Merthyr Tydfil